CLINICAL TRIAL: NCT04019925
Title: Assessing the Wear Rates of the ADM/MDM Dual Mobility Hips Manufactured by Stryker Orthopaedics Using 3D X-ray Analysis
Brief Title: Assessing the Wear Rates of the ADM/MDM Hips Using 3D X-ray Analysis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Unity Health Toronto (Other)
Collaborators: Stryker Orthopaedics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-061
Record Dates: First submitted 2019-07-03; First posted 2019-07-15 (Actual); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: Arthroplasty, Replacement, Hip

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- ADM/MDM hip prosthesis (Other): Type of prosthesis participant received.
  Interventions: Device: ADM/MDM hip

INTERVENTIONS:
Device: ADM/MDM hip — Dual Mobility Hip prosthesis manufactured by Stryker Orthopaedics: ADM/MDM
  Other Names: Dual Mobility Hip

SUMMARY:
A common complication post hip replacement is hip dislocation or hip instability which can lead to the hip implants being revised. A new generation of Dual Mobility hips was designed to minimize hip dislocation/hip instability and polyethylene wear thus increasing the longevity of the hip prosthesis and reducing the number of re-operations for a patient. In this study we will be assessing 2 dual mobility hips manufactured by Stryker Orthopaedics Inc. The ADM and the MDM.

DETAILED DESCRIPTION:
Hip replacement is a procedure in which the hip joint is replaced by a prosthetic implant or prosthesis. Post op hip dislocation or hip instability is a common complication which can lead to the hip implants being revised. There are many types of hip prostheses manufactured with the aim of prolonging longevity of the prosthesis and minimizing postoperative complications. One of these is a new generation of dual mobility hip manufactured by Stryker Orthopaedics. The Anatomic Dual Mobility (ADM) and the Modular Dual Mobility (MDM) were designed to minimize hip dislocation/hip instability and polyethylene wear thus increasing the longevity of the hip prosthesis and reducing the number of re-operations for a patient. In this study we will be assessing the outcome of the ADM and MDM hip system.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant female
* Skeletally mature
* 18 to 75 years old
* Stryker Dual Mobility Hip prosthesis
* BMI between 20 and 35
* Follow-up x-rays between 3 years and 6 years postop

Exclusion Criteria:

* Dual Mobility Hip implant that is not the ADM or MDM
* BMI that is 19 or less
* BMI that is greater than 36
* Most recent x-rays less than 3 years postop

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2020-03-30 (Estimated); Study Completion 2020-08-31 (Estimated)

PRIMARY OUTCOMES:
To assess the change in polyethylene wear of Dual Mobility hip implants using Stryker Orthopaedics ADM & MDM prostheses | before the patient's discharge home, 6 weeks postop, and the most recent x-ray taken up to 5 years postop.
  This study will assess the change in linear and volumetric wear using 3D x-ray analysis. Measurements will be taken of x-rays obtained before the patient's discharge home, 6 weeks postop, and the most recent x-ray taken more than 3 years postop.

SECONDARY OUTCOMES:
To review the number of postop hip dislocations/hip instabilities | first 5 years post surgery
  Dislocations and the post op time for each occurrence per patient will be collected in tabular format. This in turn will be used to calculate percent of cases/subject.

CONTACTS AND LOCATIONS:
Overall Officials: Amit Atrey, MD, Principal Investigator — Unity Health Toronto, St. Michael's Hospital
Locations (1):
- Unity Health Toronto, St. Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huo MH, Parvizi J, Bal BS, Mont MA. What's new in total hip arthroplasty. J Bone Joint Surg Am. 2009 Oct;91(10):2522-34. doi: 10.2106/JBJS.I.00801. No abstract available. PMID 19797590
- [Background] Barrack RL. Dislocation after total hip arthroplasty: implant design and orientation. J Am Acad Orthop Surg. 2003 Mar-Apr;11(2):89-99. doi: 10.5435/00124635-200303000-00003. PMID 12670135
- [Background] Khatod M, Barber T, Paxton E, Namba R, Fithian D. An analysis of the risk of hip dislocation with a contemporary total joint registry. Clin Orthop Relat Res. 2006 Jun;447:19-23. doi: 10.1097/01.blo.0000218752.22613.78. PMID 16741469
- [Background] Goel A, Lau EC, Ong KL, Berry DJ, Malkani AL. Dislocation rates following primary total hip arthroplasty have plateaued in the Medicare population. J Arthroplasty. 2015 May;30(5):743-6. doi: 10.1016/j.arth.2014.11.012. Epub 2014 Nov 26. PMID 25573179
- [Background] Hailer NP, Weiss RJ, Stark A, Karrholm J. The risk of revision due to dislocation after total hip arthroplasty depends on surgical approach, femoral head size, sex, and primary diagnosis. An analysis of 78,098 operations in the Swedish Hip Arthroplasty Register. Acta Orthop. 2012 Oct;83(5):442-8. doi: 10.3109/17453674.2012.733919. Epub 2012 Oct 8. PMID 23039167
- [Background] Kostensalo I, Junnila M, Virolainen P, Remes V, Matilainen M, Vahlberg T, Pulkkinen P, Eskelinen A, Makela KT. Effect of femoral head size on risk of revision for dislocation after total hip arthroplasty: a population-based analysis of 42,379 primary procedures from the Finnish Arthroplasty Register. Acta Orthop. 2013 Aug;84(4):342-7. doi: 10.3109/17453674.2013.810518. Epub 2013 Jun 25. PMID 23799348
- [Background] Philippot R, Camilleri JP, Boyer B, Adam P, Farizon F. The use of a dual-articulation acetabular cup system to prevent dislocation after primary total hip arthroplasty: analysis of 384 cases at a mean follow-up of 15 years. Int Orthop. 2009 Aug;33(4):927-32. doi: 10.1007/s00264-008-0589-9. Epub 2008 Jun 3. PMID 18521598
- [Background] Darrith B, Courtney PM, Della Valle CJ. Outcomes of dual mobility components in total hip arthroplasty: a systematic review of the literature. Bone Joint J. 2018 Jan;100-B(1):11-19. doi: 10.1302/0301-620X.100B1.BJJ-2017-0462.R1. PMID 29305445
- [Background] De Martino I, D'Apolito R, Soranoglou VG, Poultsides LA, Sculco PK, Sculco TP. Dislocation following total hip arthroplasty using dual mobility acetabular components: a systematic review. Bone Joint J. 2017 Jan;99-B(ASuppl1):18-24. doi: 10.1302/0301-620X.99B1.BJJ-2016-0398.R1. PMID 28042114
- [Background] Harwin SF, Sultan AA, Khlopas A, Chughtai M, Sodhi N, Piuzzi NS, Mont MA. Mid-Term Outcomes of Dual Mobility Acetabular Cups for Revision Total Hip Arthroplasty. J Arthroplasty. 2018 May;33(5):1494-1500. doi: 10.1016/j.arth.2017.12.008. Epub 2017 Dec 14. PMID 29307678
- [Background] Loving L, Lee RK, Herrera L, Essner AP, Nevelos JE. Wear performance evaluation of a contemporary dual mobility hip bearing using multiple hip simulator testing conditions. J Arthroplasty. 2013 Jun;28(6):1041-6. doi: 10.1016/j.arth.2012.09.011. Epub 2013 Feb 22. PMID 23434106
- [Background] D'Apuzzo MR, Koch CN, Esposito CI, Elpers ME, Wright TM, Westrich GH. Assessment of Damage on a Dual Mobility Acetabular System. J Arthroplasty. 2016 Aug;31(8):1828-35. doi: 10.1016/j.arth.2016.01.039. Epub 2016 Jan 30. PMID 26897488